CLINICAL TRIAL: NCT06483217
Title: Optimal Injection Interval for Intra-Detrusor Botulinum Toxin: A Randomized Controlled Trial Utilizing a Patient-Centered Approach
Brief Title: Optimal Injection Interval for Intra-Detrusor Botulinum Toxin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Zachary S Selzler, MD, Zachary Selzler MD, Urogynecology Fellow, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #7564
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Overactive Bladder; Urinary Urgency; Urinary Incontinence; Urge Urinary Incontinence
Keywords: intradetrusor botulinum toxin; intravesical botox; intradetrusor botox; bladder chemodenervation; botox; chemodenervation; overactive bladder; urge urinary incontinence; intravesical botulinum toxin
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Standard 6 month post-operative follow up interval for repeat injection
- Patient-directed follow up (Experimental): Post-operative follow up interval for repeat injection decided by patient based on OAB symptomatology (3-12 months)
  Interventions: Behavioral: Patient-directed follow up

INTERVENTIONS:
Behavioral: Patient-directed follow up — Patients will be instructed to follow up for repeat injection based on bladder symptomatology at their own self-determined time interval.
  Arms: Patient-directed follow up

SUMMARY:
The goal of this clinical trial is to see if patients deciding their own follow up times can increase the effectiveness of botulinum toxin (BTX or "Botox") injection for overactive bladder (OAB). The main questions it aims to answer are:

* Does the time between repeat injections differ from the 6-month standard when it is based on patient symptoms alone?
* Does symptom control or patient satisfaction change when patients control their own follow up times?

Participants will undergo standard botulinum toxin injection into the bladder for OAB treatment and will then be randomly assigned to follow up either at a standard 6-month interval or whenever they feel their symptoms return.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is defined by symptoms of urinary urgency, frequency, or nocturia with or without incontinence in the absence of urinary tract infection or other attributable pathology. This disease affects up to 40% of women in the United States and can have a significant impact on quality of life. It is expected to increase in prevalence with the aging US population. There are a wide variety of treatment options for OAB which range from fluid management and lifestyle modifications (first line therapy), pelvic floor physical therapy and oral medications (second line therapy), and procedural interventions such as neuromodulation or intravesical botulinum toxin (BTX-A) injections (third line therapy).

BTX-A is a potent neurotoxin derived from the anaerobic bacterium Clostridium botulinum that inhibits presynaptic release of acetylcholine from motor neurons at the neuromuscular junction to induce flaccid paralysis of musculature. It has also been found to affect sensory responses of nerve afferent nerve fibers and likely has a complex multifactorial effect on the release of excitatory neurotransmitters. Because of this, injection of BTX-A into the detrusor muscle of the bladder has become a highly effective treatment option for OAB, first approved by the FDA in January 2013. Prior studies have demonstrated superior efficacy of intravesical BTX-A injections compared to anticholinergic medication and a greater reduction in urge urinary incontinence episodes than sacral neuromodulation.

The effect of intravesical BTX-A is temporary due to turnover of presynaptic molecules. Typical chemodenervation of muscular tissue lasts 3 to 6 months based on histologic evidence, however this does not translate directly to duration of OAB symptom control given the gradual nature of neurotransmitter repletion. The largest prior trial of intravesical BTX-A demonstrated a median interval of 350 days between first and second injection, but other studies have shown a wide range of duration from 5 to 15 months. The current FDA recommendation for repeat injection is to be "considered when the clinical effect from the previous injection has diminished" with a median interval in their double-blinded placebo-controlled studies of 169 days.

Despite this recommendation, there is a wide variety in practice patterns for repeat injections, including the use of a "one size fits all" approach with standardized repeat injections at 6-month intervals. Combined with varying rates of tolerability and treatment failure, this has resulted in inconsistent data on continuation and dropout rates for repeat injections, with reported continuation rates of 20-60% in different studies. Additionally, no prior studies have reported whether repeat injection intervals have been provider- or patient-determined, nor with data on patient satisfaction ratings. Further studies are needed to better delineate optimal injection interval as well as incorporate data on what methods lead to the highest patient satisfaction and symptom control.

The purpose of this study is to ascertain the optimal time interval to repeat injection will be when it is purely patient directed based on symptomatology. Investigators will also evaluate patient satisfaction with this approach compared to standardized repeat injection interval of six months. This has the potential to change the way OAB is managed by allowing patients to control the interval to repeat injection in a safe and controlled manner. Investigators hypothesize that a patient-centered approach to repeating BTX-A injections will be similar to the standard FDA 6-month interval while leading to higher patient satisfaction and continuation rates without compromising safety or efficacy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of overactive bladder, detrusor overactivity, urinary urgency, urinary frequency, nocturnal polyuria, or urge urinary incontinence
* pursuing treatment with intravesical botulinum toxin injections

Exclusion Criteria:

- non-OAB diagnosis such as pelvic pain or interstitial cystitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Injection interval | Days from initial injection to repeat injection, up to 365 days
  time to repeat injection (days)

SECONDARY OUTCOMES:
Patient Satisfaction | 1-2 weeks post-injection
  Scores from the Surgical Satisfaction Questionnaire (SSQ-8), which contains 8 questions on satisfaction with a likert scale rating of 1-5. Higher scores indicate higher patient satisfaction.
Symptom Control | baseline scores immediately pre-injection, post-treatment scores 1-2 weeks post-injection
  Scores from the Overactive Bladder Assessment Tool (OAB-Q), which contains 5 questions on symptoms and 5 questions on quality of life with a likert scale rating of 0-5. Higher scores on the symptom section indicate WORSE overactive bladder symptoms and higher scores on the quality of life section indicate higher levels of bother/WORSE quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Peacock, MD, Principal Investigator — Louisiana State University Health Science Center - New Orleans
Locations (1):
- Louisiana State University Health Science Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] de Groat WC, Yoshimura N. Afferent nerve regulation of bladder function in health and disease. Handb Exp Pharmacol. 2009;(194):91-138. doi: 10.1007/978-3-540-79090-7_4. PMID 19655106
- [Background] Amundsen CL, Richter HE, Menefee SA, Komesu YM, Arya LA, Gregory WT, Myers DL, Zyczynski HM, Vasavada S, Nolen TL, Wallace D, Meikle SF. OnabotulinumtoxinA vs Sacral Neuromodulation on Refractory Urgency Urinary Incontinence in Women: A Randomized Clinical Trial. JAMA. 2016 Oct 4;316(13):1366-1374. doi: 10.1001/jama.2016.14617. PMID 27701661
- [Background] Amundsen CL, Komesu YM, Chermansky C, Gregory WT, Myers DL, Honeycutt EF, Vasavada SP, Nguyen JN, Wilson TS, Harvie HS, Wallace D; Pelvic Floor Disorders Network. Two-Year Outcomes of Sacral Neuromodulation Versus OnabotulinumtoxinA for Refractory Urgency Urinary Incontinence: A Randomized Trial. Eur Urol. 2018 Jul;74(1):66-73. doi: 10.1016/j.eururo.2018.02.011. Epub 2018 Feb 24. PMID 29482936
- [Background] Granese R, Adile G, Gugliotta G, Cucinella G, Saitta S, Adile B. Botox((R)) for idiopathic overactive bladder: efficacy, duration and safety. Effectiveness of subsequent injection. Arch Gynecol Obstet. 2012 Oct;286(4):923-9. doi: 10.1007/s00404-012-2349-8. Epub 2012 May 24. PMID 22622849
- [Background] Dowson C, Watkins J, Khan MS, Dasgupta P, Sahai A. Repeated botulinum toxin type A injections for refractory overactive bladder: medium-term outcomes, safety profile, and discontinuation rates. Eur Urol. 2012 Apr;61(4):834-9. doi: 10.1016/j.eururo.2011.12.011. Epub 2011 Dec 13. PMID 22204745
- See also: FDA Medication Guide for onabotulinumtoxinA, accessed June 28th 2024 — https://www.accessdata.fda.gov/drugsatfda_docs/label/2023/103000s5327lbl.pdf